CLINICAL TRIAL: NCT01960803
Title: Lumpectomy Followed By Intraoperative Electron Radiation Therapy (IOERT) As A Single, Full Dose Partial Breast Irradiation For Early Stage, Node Negative, Invasive Breast Cancer
Brief Title: Lumpectomy Followed By Intraoperative Electron Radiation Therapy (IOERT)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IOERT is no longer an experimental treatment and was now offered as SOC to patients experiencing IBC. As this therapy is being offered to them regardless of study participation at numerous institutions across the country.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACI-001
Record Dates: First submitted 2013-09-25; First posted 2013-10-11 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Invasive Ductal Breast Cancer; Carcinoma Breast Stage I
Keywords: Stage I Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IOERT arm (Experimental): Intraoperative electron radiotherapy (IOERT) is delivered after completion of the lumpectomy and sentinel node procedure. IOERT is performed on a mobile self-shielded magnetron-driven X-band linear accelerator specifically developed for use in the operating room. This machine produces megavoltage electron beams of energy ranging between 4 and 12 MeV. The radiation is delivered from the device to the tumor bed through an attached applicator. A single dose of 21 Gy calculated to the 90% depth posterior to the tumor bed will be administered and will last approximately 2.5 minutes.
  Interventions: Radiation: Intraoperative Electron Radiotherapy

INTERVENTIONS:
Radiation: Intraoperative Electron Radiotherapy — Intraoperative Electron Radiotherapy (IOERT) is delivered after completion of the lumpectomy and sentinel node procedure.

SUMMARY:
The overall objective of this study is to determine the feasibility and tolerability of single dose Intraoperative Electron Radiation Treatment ("IOERT") as definitive therapy when administered at the time of breast conserving surgery for patients with early stage breast cancer.

DETAILED DESCRIPTION:
Evaluate local and distant recurrence rates and cosmetic outcomes. Both clinical evaluation of cosmetic outcome by the Surgeon, and subjective impression of cosmetic outcome by the patient, are evaluated using questionnaire.

Local recurrence is evaluated under the same imaging protocol used for Whole breast radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patient agrees to breast conservation therapy (segmental resection, partial mastectomy, and radiation therapy) as the treatment for their breast cancer
* Patient agrees to evaluation of the axilla with sentinel lymph node biopsy
* Peri or post-menopausal women age > 50, defined as women who have experienced no menstrual period in the past 6 months or more
* BRCA1 and 2 gene mutation negative, if tested. [genetic testing is NOT required based upon personal or family history]
* Unifocal (unicentric), invasive ductal carcinoma or favorable sub-types (mucinous, tubular, colloid) < 2.0 cm in diameter, primary T-stage of Tis or T1 (AJCC criteria)
* Grade 1, 2, or 3 acceptable
* Associated LCIS is allowed
* Pure DCIS allowed if <2.5 cm, low to intermediate nuclear grade and resected margins negative at > 3 mm (per ASTRO criteria)
* Estrogen receptor (ER) status of positive
* Patient has clear margins >2 mm on gross pathologic examination
* Patient is node-negative, defined as N0 (i-) or N0 (i+)
* Patient must be deemed functionally and mentally competent to understand and sign the informed consent
* Neoadjuvant hormonal therapy is allowed if all other ASTRO suitable criteria have been met prior to onset of hormonal therapy

Exclusion Criteria:

* Prior breast malignancy or other malignancy if metastatic, or with expected survival of < 5 years
* Immunocompromised status
* Pregnancy
* Women with an active connective tissue disorder (i.e. scleroderma, lupus and others)
* Breast cancer that involves the skin or chest wall, locally advanced breast cancer
* Invasive lobular carcinoma
* Evidence of lymphovascular invasion (LVI)
* Invasive carcinoma with extensive intraductal component (EIC)
* Neoadjuvant chemotherapy
* Patients with 1 or more positive lymph node determined during surgery with sentinel node and/or axillary dissection
* Someone who is not a candidate for breast conserving management, i.e., prior whole breast radiation therapy

Ages: 50 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
To evaluate change over time on the incidence of local and distance recurrence rates. | 1 month, 3 months, 6 months, 12 months, and then annually for 10 years.
  Subjects will be followed for recurrence rates at one month, three months, six months, twelve months, and then annually for up to 10 years. This will include: history and physical exam, as well as radiographic images at physician discretion and per study protocol.

SECONDARY OUTCOMES:
To evaluate changes in the short-term and long-term side effects related to IOERT | 1 month, 3 months, 6 months, 12 months, and then annually for 10 years.
  Assessment of the overall patient satisfaction related to the therapy and cosmetic outcome. Cosmesis will be scored by both the physician and patient using the RTOG cosmesis rating system at one month, three months, six months, twelve months, and 24 months. The secondary outcome measure will only take place in the first two years of the 10 year time frame for patient follow up. After 24 month evaluations, patients will only be followed for incidence of local and distance recurrence rates.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Krueger, MD FACS, Principal Investigator — Advocate Health Care - Advocate Christ Medical Center
Locations (1):
- Advocate Christ Medical Center, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No